CLINICAL TRIAL: NCT05800782
Title: Examining the Effectiveness of Face Perception and Memory Training to Improve Face Recognition in Developmental Prosopagnosia
Brief Title: Face Perception vs. Memory Training to Improve Face Recognition in Developmental Prosopagnosia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston VA Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01EY032510-02 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-04-06 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-03

CONDITIONS: Developmental Prosopagnosia
MeSH Terms: conditions — Prosopagnosia

STUDY DESIGN:
Intervention Model Description: There will be a pre assessment, 6 weeks of training/active control, then an immediate post assessment, and finally an assessment after a 12-week no-contact period
Who Masked: Participant
Masking Description: Participants will not be told whether they are in the experimental or control conditions and all conditions will require discriminating faces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Memory Training (Experimental): Participants will perform 6 weeks of face memory training (5 x 40 min sessions/week) that targets enhancing encoding to improve face recollection. As training progresses, the repetition lags (spaces between repeated foil faces) and number of faces will increase.
  Interventions: Behavioral: Face Memory Training
- Perception Training (Active Comparator): Participants will perform 6 weeks of face perception training (5 x 40 min sessions/week) that require discriminating faces based on internal features (e.g., eyebrow-eye distance). As training progresses, the faces will become more challenging and the face sizes will vary.
  Interventions: Behavioral: Face Perception Training
- Active Control Training (Placebo Comparator): Participants will perform 6 weeks of face perception training (5 x 40 min sessions/week) that require discriminating faces based on external facial features (e.g., hair). As training progresses, the faces will become more challenging and the face sizes will vary.
  Interventions: Behavioral: Placebo control training

INTERVENTIONS:
Behavioral: Face Memory Training — Computer-based training using faces targeting face memory
  Arms: Memory Training
Behavioral: Face Perception Training — Computer-based training using faces targeting improving face perception
  Arms: Perception Training
Behavioral: Placebo control training — Computer-based training using faces not targeting improving face perception or memory
  Arms: Active Control Training

SUMMARY:
The goal of this study is to test the effectiveness of two experimental training programs aimed at improving face processing in developmental prosopagnosia (perception training, memory training) in comparison to an active control. The investigators will use a longitudinal design and randomize developmental prosopagnosics to three parallel arms: active control, perception training and memory training.

DETAILED DESCRIPTION:
The investigators propose a longitudinal design with three parallel arms: active control, perception training and memory training. To maximize power, developmental prosopagnosics (DPs) in the active control group will be subsequently be offered training. Pre-training/control assessments will be performed and within 2 weeks, DPs will be randomized to one of the three training conditions. Next, all DPs will complete 6-weeks of their assigned intervention. The research assistant will provide coaching at least once per week. DPs will be assessed within two weeks of training completion and after a 12-week no-contact period. For those in the active control group, the no-contact period will serve to wash out any placebo effect and Assessment 3 will be used as their new baseline. These DPs will then be randomized to perception or memory training. Assessments will then be given to these DPs within a week after intervention completion and after a 12 weeks no-contact period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90
* Have lifelong histories of face recognition difficulties that impact everyday life (i.e., not associated with some event such as a stroke, seizure, etc)
* Score > 2 standard deviations below the mean on the famous faces test and Cambridge Face Memory Test. This is in line with our previous studies and others in the literature.

Exclusion Criteria:

* History of a significant neurological disorder including hydrocephalus, stroke, moderate to severe traumatic brain injury (TBI), severe neuromuscular diseases, or severe hypoxia due to cardiac arrest.
* Participants with a history of mild TBI or simple concussion will not be excluded as long as it was > 6 months ago and as long as they have not had repeated concussions (>5).
* Participants will be excluded if they have impairments that interfere with cognitive performance, such as uncorrected hearing or vision, lack of English proficiency, musculoskeletal or other issues.
* Additionally, participants will be excluded if they have psychiatric disorders, such as schizophrenia, major depressive disorder, bipolar disorder, chronic intractable obsessive-compulsive disorder, or agoraphobia.
* Participants with a diagnosis of ADHD will be included as long as their medication has been consistent for the past 6 months.
* Participants who are currently dependent on alcohol or other substances will be excluded, as this may negatively impact cognitive performance.
* Participants who currently are, or within the last 6 months, participating in a behavioral or pharmacological intervention will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in Cambridge Face Memory Test from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  unfamiliar face learning/memory test, Cambridge Face Memory Test, minimum=0/maximum=72, higher is better performance
Change in Face Perception from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  computerized Benton Face Recognition Test, minimum=0/maximum=54, higher is better performance

SECONDARY OUTCOMES:
Change in Face Recollection from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  face recollection measure derived from old/new unfamiliar face recognition test
Change in Self-reported face recognition ability from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline),12 weeks after training ends (approximately 22 weeks after baseline)
  items assessing everyday face recognition, minimum=0/maximum=100, higher is better
Change in Eye processing ability from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  average eye processing ability from Georges task
Change in Holistic processing from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  measure of holistic processing of faces (holistic advantage) from part-whole task
Change in NIH PROMIS Social functioning self-report from baseline to post-training | baseline, within 2 weeks post-training (approximately 10 weeks after baseline), 12 weeks after training ends (approximately 22 weeks after baseline)
  bank of NIH PROMIS items asking about social functioning related to prosopagnosia, minimum=0/maximum=100, higher is better

CONTACTS AND LOCATIONS:
Overall Officials: Joseph DeGutis, Ph.D., Principal Investigator — Harvard Medical School/VA Boston Healthcare Systems
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to other researchers in accordance with the VA Boston Healthcare System IRB and Privacy/Security policies
Supporting Information: CSR, Analytic Code
Time Frame: Once the VA Boston Healthcare System IRB approves sharing this information
Access Criteria: The VA Boston Healthcare System IRB will also establish access criteria